CLINICAL TRIAL: NCT06475872
Title: Open, Randomized, 2-Group, 2-Period, Fasting, Single-Dose, Crossover Study to Evaluate the Bioequivalence of "Crecheck Tablet 2.5 mg (Rosuvastatin Calcium)" of Hanlim Pharm. Co., Ltd. and "Crestor Tablet 5 mg (Rosuvastatin Calcium)" of AstraZeneca Korea Co., Ltd. in Healthy Adult Subjects
Brief Title: Study to Evaluate the Bioequivalence of "Crecheck Tablet 2.5 mg (Rosuvastatin Calcium)" and "Crestor Tablet 5 mg (Rosuvastatin Calcium)" in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KMRI-BE-23021
Record Dates: First submitted 2024-06-17; First posted 2024-06-26 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Primary Hypercholesterolemia; Combined Hyperlipidemia
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crecheck Tab (Experimental): On the day of the visit, take 2 tablets of the test drug orally with 150 mL of water around 8 am.
  Interventions: Drug: Crecheck Tablet 2.5 mg
- Comparator (Active Comparator): On the day of the visit, take 1 tablet of the comparator drug orally with 150 mL of water around 8 am.
  Interventions: Drug: Crestor Tablet 5 mg

INTERVENTIONS:
Drug: Crecheck Tablet 2.5 mg — 2 tablets orally once a day
  Other Names: Rosuvastatin Calcium
  Arms: Crecheck Tab
Drug: Crestor Tablet 5 mg — 1 tablet orally once a day
  Other Names: Rosuvastatin Calcium
  Arms: Comparator

SUMMARY:
This clinical trial is an open, randomized, 2-group, 2-period, fasting, single-dose, crossover study to evaluate the bioequivalence of "Crecheck Tablet 2.5 mg (Rosuvastatin Calcium)" of Hanlim Pharm. Co., Ltd. and "Crestor Tablet 5 mg (Rosuvastatin Calcium)" of AstraZeneca Korea Co., Ltd. in healthy adult subjects.

DETAILED DESCRIPTION:
This study is to compare and evaluate the safety and pharmacokinetic characteristics of Hanlim Pharm. Co., Ltd.'s "Crecheck Tablet 2.5 mg (Rosuvastatin Calcium)" as the test drug and AstraZeneca Korea Co., Ltd.'s "Crestor Tablet 5 mg (Rosuvastatin Calcium)" as the reference drug in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 years or older at the time of screening
2. Individuals with no clinically significant congenital or chronic diseases and no pathological symptoms or findings based on medical examinations (such as EEG, ECG, chest and gastric endoscopy, or gastrointestinal radiology tests, if necessary)
3. Individuals deemed suitable for the study based on screening tests (e.g., hematology, blood chemistry, serology, and urinalysis) as determined by the principal investigator (or a designated sub-investigator)
4. Individuals with a Body Mass Index (BMI) between 18.0 and 30.0 (BMI calculation: weight (kg) / height (m)²)
5. Individuals who have received and understood a thorough explanation of the study's purpose, content, investigational drug characteristics, and potential adverse events, and have voluntarily decided to participate and agreed in writing to comply with the study requirements during the trial period
6. Individuals who agree to use medically recognized contraceptive methods* (excluding hormonal contraceptives) to avoid pregnancy from the first administration of the investigational drug until one week after the last administration * Medically recognized contraceptive methods: intrauterine devices (IUD, IUS), vasectomy, tubal ligation, and combined barrier methods (male condoms, female condoms, cervical caps, diaphragms, sponges, etc.), or if using spermicides, combined use of two or more barrier methods

Exclusion Criteria:

1. Individuals who have taken enzyme-inducing or inhibiting drugs such as barbiturates within 30 days before the start of the study (first dosing day) or medications that might interfere with the study within 10 days before the start of the study (first dosing day)
2. Individuals who have engaged in excessive alcohol consumption within one month before the start of the study (first dosing day)

   * For men, more than an average of 21 drinks per week
   * For women, more than an average of 14 drinks per week (One drink: 45 mL of distilled spirits or 360 mL of beer or 150 mL of wine)
3. Individuals who have participated in clinical trials (including bioequivalence studies) and received investigational drugs within six months before the start of the study (first dosing day)
4. Individuals who have donated whole blood within 8 weeks or donated blood components within 2 weeks before the start of the study (first dosing day)
5. Individuals with a history of gastrointestinal surgery that may affect drug absorption
6. Patients with the following conditions:

   * Hypersensitivity to the components of this drug
   * Active liver disease, including unexplained persistent elevations in serum transaminases or serum transaminase levels exceeding three times the upper limit of normal
   * Myopathy
   * Concurrent use of cyclosporine
   * Severe renal impairment (creatinine clearance (CLcr) < 30 mL/min)
   * Pregnant or lactating women, and women of childbearing potential not using adequate contraceptive methods
   * Patients prone to myopathy/rhabdomyolysis (contraindicated when administered at a 40 mg dose of this drug)
   * Moderate renal impairment (creatinine clearance < 60 mL/min)
   * Hypothyroidism
   * A history or family history of hereditary muscle disorders
   * A history of muscle toxicity with other HMG-CoA reductase inhibitors or fibrates
   * Alcoholism
   * Situations where plasma concentrations may increase
   * Asian patients
   * Concurrent use of fibrates
   * Genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, since this product contains lactose
7. Individuals with a history of mental illness
8. Individuals deemed unsuitable for this clinical trial for reasons other than the above inclusion/exclusion criteria by the principal investigator (or a designated sub-investigator)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 48 hours
  Concentration of rosuvastatin in plasma
Peak Plasma Concentration (Cmax) | 48 hours
  Concentration of rosuvastatin in plasma

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration (Tmax) | 48 hours
  Concentration of rosuvastatin in plasma
Half Life (t1/2) | 48 hours
  Concentration of rosuvastatin in plasma
AUC∞ | 48 hours
  Concentration of rosuvastatin in plasma
AUCt/AUC∞(%) | 48 hours
  Concentration of rosuvastatin in plasma
Dissolution pattern by comparative dissolution test of Rosuvastatin | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seok Gyeong Medical Foundation Central Hospital, Gyeonggi-do, South Korea